CLINICAL TRIAL: NCT03504852
Title: A Randomized, Double-blind, Multicenter Study Assessing Short and Long-term Efficacy, Safety, and Tolerability of Sub-cutaneous Secukinumab in Subjects of Body Weight 90 kg or Higher With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Efficacy and Safety of 2 Secukinumab Regimens in 90kg or More Weight Group With Moderate/Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CAIN457A2324; 2015-004620-60 (EudraCT Number)
Record Dates: First submitted 2018-03-29; First posted 2018-04-20 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Moderate to Severe Chronic Plaque-type Psoriasis
Keywords: psoriasis; secukinumab; immune-mediated systemic disease; papules; plaques; itching; weight
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid; Pruritus; Body Weight | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab 300 mg every 2 weeks (Q2W) (Experimental): 2 injections of secukinumab 150 mg once weekly up to week 4 and thereafter every 2 weeks. Subjects remained on secukinumab 300 mg every 2 weeks until the end of treatment.
  Interventions: Drug: secukinumab 150 mg
- Secukinumab 300 mg every 4 weeks (Q4W) (Active Comparator): 2 injections of secukinumab 150 mg once weekly up to week 4 and thereafter Q4W. Includes both subjects randomized to remain on Q4W the entire treatment period, and subjects that were Psoriasis Area and Severity Index (PASI) 90 responders at Week 16 from the secukinumab 300 mg Q4W possible up-titrate group.
  Interventions: Drug: secukinumab 150 mg
- Secukinumab 300 mg every 4 weeks non-responders up-titration (Q4W NR up) (Active Comparator): 2 injections of secukinumab 150 mg once weekly up to week 4, then Q4W up to Week 16 and thereafter Q2W. Includes Psoriasis Area and Severity Index (PASI) 90 non-responders (NR) at Week 16 from the secukinumab 300 mg Q4W possible up-titrate group (subjects randomized to switch to Q2W if PASI 90 non-responder at Week 16).
  Interventions: Drug: secukinumab 150 mg

INTERVENTIONS:
Drug: secukinumab 150 mg — sub-cutaneous secukinumab prefilled syringe 150 mg

SUMMARY:
The purpose of this study is to assess secukinumab high dose (every 2 weeks) vs standard dose (every 4 weeks) in heavy body weight subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
A 52-week multicenter, randomized, double-blind, parallel-group trial in 331 subjects with moderate to severe chronic plaque-type psoriasis of body weight 90 kg or higher at time of randomization.

This study consisted of 4 periods: screening (up to 4 weeks), treatment Period 1 (16 weeks), treatment Period 2 (36 weeks), and post-treatment follow-up (8 weeks).

Subjects were randomized using a 1:1 ratio to the following groups: Secukinumab 300 mg every 2 weeks; Secukinumab 300 mg every 4 weeks.

In addition, subjects from the 300 mg every 4 weeks group who did not achieve Psoriasis Area Severity Index (PASI) 90 response at Week 16 were reassigned using a 1:1 ratio to either remain on secukinumab 300 mg every 4 weeks or receive secukinumab 300 mg every 2 weeks starting at Week 16, until the end of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent must have been obtained before any assessment was performed. Where relevant, a legal representative will also have signed the informed study consent according to local laws and regulations.
* Subjects must have been able to understand and communicate with the investigator and comply with the requirements of the study.
* Men or women at least 18 years of age at time of screening.
* Body weight of ≥ 90 kg at the time of randomization.
* Chronic plaque-type psoriasis present for at least 6 months and diagnosed before randomization.
* Moderate to severe psoriasis as defined at randomization by:

  * Psoriasis Area and Severity Index (PASI) score of 12 or greater, and
  * Investigator's Global Assessment (IGA) mod 2011 score of 3 or greater (based on a static scale of 0 - 4), and
  * Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater.
* Candidate for systemic therapy. This is defined as a subject having moderate to severe chronic plaque-type psoriasis that is inadequately controlled by:

  * topical treatment and/or,
  * phototherapy and/or,
  * previous systemic therapy.

Key Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at screening or Randomization.
* Ongoing use of prohibited treatments. Washout periods detailed in the protocol have to be adhered to. Subjects not willing to limit ultraviolet (UV) light exposure (e.g., sunbathing and / or the use of tanning devices) during the course of the study will be considered not eligible for this study since UV light exposure is prohibited. Note: administration of live vaccines 6 weeks prior to Randomization or during the study period is also prohibited.
* Previous exposure to secukinumab (AIN457) or any other biologic drug directly targeting Interleukin-17 (IL-17) or the IL-17 receptor.
* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 4 weeks until the expected pharmacodynamic effect has returned to baseline, whichever is longer; or longer if required by local regulations.
* Pregnant or nursing (lactating) women
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for skin Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
* History of hypersensitivity to any of the study drug constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (65):
- United States (37):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Rogers, Arkansas
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Centennial, Colorado
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Alpharetta, Georgia
  - Novartis Investigative Site, Snellville, Georgia
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, New Albany, Indiana
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New Brighton, Minnesota
  - Novartis Investigative Site, Saint Joseph, Missouri
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, Forest Hills, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Fairborn, Ohio
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Pflugerville, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Wenatchee, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- Canada (6):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Red Deer, Alberta
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Guelph, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Québec
- Czechia (2):
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Nový Jičín
- Germany (5):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
- Hungary (3):
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Italy (5):
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Napoli
- Russia (7):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Lipetsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Augustin M, Reich K, Yamauchi P, Pinter A, Bagel J, Dahale S, You R, Bruin G, Djimopoulos J, Paguet B, Charef P, Patekar M, Keefe D. Secukinumab dosing every 2 weeks demonstrated superior efficacy compared with dosing every 4 weeks in patients with psoriasis weighing 90 kg or more: results of a randomized controlled trial. Br J Dermatol. 2022 Jun;186(6):942-954. doi: 10.1111/bjd.20971. Epub 2022 Apr 8. PMID 34981829
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=862

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 331 participants in the study were randomized and 330 participants were treated. (One participant in the Secukinumab 300 mg Q4W arm was randomized but not treated. This participant was included in the randomization (demographic and disposition) set and the full analysis set, but was not included in the safety (Adverse Events) set.)
Groups:
- Secukinumab 300 mg Every 4 Weeks (Q4W) (Safety): 2 injections of secukinumab 150 mg once weekly up to week 4 and thereafter Q4W. Includes both subjects randomized to remain on Q4W the entire treatment period, and subjects that were Psoriasis Area and Severity Index (PASI) 90 responders at Week 16 from the secukinumab 300 mg Q4W possible up-titrate group.
Period: Overall Study
Arm/Group | Secukinumab 300 mg Every 2 Weeks (Q2W) | Secukinumab 300 mg Every 4 Weeks (Q4W) (Safety) | Secukinumab 300 mg Every 4 Weeks Non-responders Up-titration (Q4W NR up)
Started | 165 | 135 | 31
Completed | 148 | 117 | 28
Not Completed | 17 | 18 | 3
Not completed — Withdrawal of informed consent | 2 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 1
Not completed — Lost to Follow-up | 4 | 1 | 0
Not completed — New therapy for study indication | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Adverse Event | 4 | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg Every 2 Weeks (Q2W) | Secukinumab 300 mg Every 4 Weeks (Q4W) (Safety) | Secukinumab 300 mg Every 4 Weeks Non-responders Up-titration (Q4W NR up) | Total
Number analyzed (Participants) | 165 | 135 | 31 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (12.73) | 46.1 (13.24) | 44.7 (13.61) | 47.1 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 34 | 10 | 83
  Male | 126 | 101 | 21 | 248
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 4 | 4 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 7 | 5 | 0 | 12
  White | 151 | 125 | 30 | 306
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieve 90% or Greater Reduction in Psoriasis Area and Severity Index (PASI) Score - Week 16 (Full Analysis Set)
Description: A subject was considered as a PASI 90 responder if s/he achieved a reduction of 90% or more of the PASI score, compared to baseline, at a given time point.The head, trunk, upper limbs and lower limbs were assessed separately for erythema, thickening, and scaling. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0, i.e., higher scores represent more severity.
Time Frame: 16 weeks
Population: Full analysis set. Please note that the Secukinumab 300 mg every 4 weeks non-responders up-titration (Q4W NR up) arm did not apply to this efficacy outcome measure and therefore no results are reported here for this arm.
Measure: Count of Participants; unit: Participants
Groups:
- Secukinumab 300 mg Every 4 Weeks (Q4W) (up to Week 16 Pre-dose): Subjects received 2 injections of secukinumab 150 mg once weekly for four weeks (at Randomization, Weeks 1, 2 and 3), followed by 2 injections of secukinumab 150 mg every four weeks, starting at Week 4 and up to Week 12.
Arm/Group | Secukinumab 300 mg Every 2 Weeks (Q2W) | Secukinumab 300 mg Every 4 Weeks (Q4W) (up to Week 16 Pre-dose)
Number analyzed (Participants) | 165 | 166
Participants | 121 | 92
Statistical Analysis 1: Comparison: Secukinumab 300 mg Every 2 Weeks (Q2W) vs Secukinumab 300 mg Every 4 Weeks (Q4W) (up to Week 16 Pre-dose); Test type: Superiority; p = 0.0003, Regression, Logistic — One-sided p-value; Risk Difference (RD) = 17.72, 95% CI 2-sided [7.45 to 27.98]
Statistical Analysis 2: Comparison: Secukinumab 300 mg Every 2 Weeks (Q2W) vs Secukinumab 300 mg Every 4 Weeks (Q4W) (up to Week 16 Pre-dose); Test type: Superiority; p = 0.0003, Regression, Logistic — One-sided p-value; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.44 to 3.78]

2. Secondary Outcome: Percentage of Subjects Who Achieve Investigator Global Assessment (IGA Modified 2011) Score of 0 or 1 - Week 16 (Full Analysis Set)
Description: IGA mod 2011 was conducted for overall psoriatic disease. The IGA modified 2011 used in this study was static, i.e., it referred exclusively to the subject's disease state at the time of the assessments, and did not attempt a comparison with any of the subject's previous disease states, whether at baseline or at a previous visit. The scale has 0 (clear) as min and 4 (severe) as max, i.e., a higher score indicates more severity.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg Every 2 Weeks (Q2W) | Secukinumab 300 mg Every 4 Weeks (Q4W) (up to Week 16 Pre-dose)
Number analyzed (Participants) | 165 | 166
Participants | 122 | 109
Statistical Analysis 1: Comparison: Secukinumab 300 mg Every 2 Weeks (Q2W) vs Secukinumab 300 mg Every 4 Weeks (Q4W) (up to Week 16 Pre-dose); Test type: Superiority; p = 0.0498, Regression, Logistic — One-sided p-value; Risk Difference (RD) = 8.28, 95% CI 2-sided [-1.65 to 18.20]
Statistical Analysis 2: Comparison: Secukinumab 300 mg Every 2 Weeks (Q2W) vs Secukinumab 300 mg Every 4 Weeks (Q4W) (up to Week 16 Pre-dose); Test type: Superiority; p = 0.0498, Regression, Logistic — One-sided p-value; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.92 to 2.47]

3. Secondary Outcome: Absolute and Relative Frequencies for Deaths, Other Serious or Clinically Significant Adverse Events or Related Discontinuations - Entire Study Period (Safety Set)
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study until the end of study visit. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 8 weeks post treatment, up to a maximum timeframe of 470 days.
Population: safety set - includes the results for the Secukinumab 300 mg every 4 weeks non-responders up-titration (Q4W NR up) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg Every 2 Weeks (Q2W) | Secukinumab 300 mg Every 4 Weeks (Q4W) (Safety) | Secukinumab 300 mg Every 4 Weeks Non-responders Up-titration (Q4W NR up)
Number analyzed (Participants) | 165 | 134 | 31
Participants
  Patients with any AE(s) | 127 | 97 | 24
  Patients with serious or other significant events - Death | 0 | 1 | 0
  Patients with serious or other significant events - Non-fatal SAE(s) | 14 | 17 | 4
  Patients with serious or other significant events - Discontinued study treatment due to any AE(s) | 4 | 9 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 8 weeks post treatment, up to a maximum timeframe of 470 days.
Groups:
- All Patients: All Patients
Arm/Group | Secukinumab 300 mg Every 2 Weeks (Q2W) | Secukinumab 300 mg Every 4 Weeks (Q4W) (Safety) | Secukinumab 300 mg Every 4 Weeks Non-responders Up-titration (Q4W NR up) | All Patients
All-Cause Mortality (participants affected / at risk) | 0/165 | 1/134 | 0/31 | 1/330
Serious Adverse Events (participants affected / at risk) | 14/165 | 18/134 | 4/31 | 36/330
Other Adverse Events (participants affected / at risk) | 66/165 | 57/134 | 16/31 | 139/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg Every 2 Weeks (Q2W) (N=165) | Secukinumab 300 mg Every 4 Weeks (Q4W) (Safety) (N=134) | Secukinumab 300 mg Every 4 Weeks Non-responders Up-titration (Q4W NR up) (N=31) | All Patients (N=330)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 2
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholestatic liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Acute HIV infection (Infections and infestations) | 0 | 1 | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 1
Blast injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Quadriplegia (Nervous system disorders) | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg Every 2 Weeks (Q2W) (N=165) | Secukinumab 300 mg Every 4 Weeks (Q4W) (Safety) (N=134) | Secukinumab 300 mg Every 4 Weeks Non-responders Up-titration (Q4W NR up) (N=31) | All Patients (N=330)
Diarrhoea (Gastrointestinal disorders) | 10 | 6 | 2 | 18
Nausea (Gastrointestinal disorders) | 1 | 4 | 2 | 7
Fatigue (General disorders) | 4 | 3 | 2 | 9
Pyrexia (General disorders) | 2 | 2 | 2 | 6
Nasopharyngitis (Infections and infestations) | 32 | 22 | 5 | 59
Tooth abscess (Infections and infestations) | 1 | 0 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 12 | 9 | 3 | 24
Urinary tract infection (Infections and infestations) | 1 | 5 | 2 | 8
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 3
Neutrophil count decreased (Investigations) | 1 | 3 | 3 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 2 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2 | 11
Headache (Nervous system disorders) | 11 | 6 | 1 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 2 | 12
Intertrigo (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03504852/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03504852/SAP_001.pdf